CLINICAL TRIAL: NCT02558595
Title: Randomized, Controlled Pilot Study of Niacinamide in Polycystic Kidney Disease
Brief Title: Pilot Study of Niacinamide in Polycystic Kidney Disease (NIAC-PKD2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alan Yu, MB, BChir, Professor of Medicine, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00002827; R21DK104086 (NIH)
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Polycystic Kidney Disease
Keywords: PKD; Kidney disease; Vitamin B3
MeSH Terms: conditions — Polycystic Kidney Diseases; Kidney Diseases | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Niacinamide (Experimental): Participants will be asked to take niacinamide at a dose of 30 mg/kg/d orally.
  Interventions: Dietary Supplement: Niacinamide
- Placebo (Placebo Comparator): Participants will be asked to take a placebo pill at a dose of 30 mg/kg/d orally.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Niacinamide
  Other Names: Nicotinamide; Vitamin B3
  Arms: Niacinamide
Other: Placebo — Placebo pill that matches niacinamide pill is size, shape and color
  Arms: Placebo

SUMMARY:
The purpose of this study is to observe the effects of niacinamide on markers of kidney injury, inflammation, kidney cyst growth and kidney function.

DETAILED DESCRIPTION:
Polycystic Kidney Disease (PKD) is a genetic disease that affects about 1 in 500 people worldwide. It can lead to kidney failure which can lead to death. PKD causes the development of kidney cysts (fluid-filled balloons), which cause worsening kidney function. It is common for people with PKD to also have blood in the urine, kidney pain, high blood pressure, kidney stones, kidney infections, and cysts in the brain or other parts of the body.

There is currently no treatment known to stop cyst growth or a cure for the disease.

Participants in this study will be randomly assigned to one of two groups: niacinamide or placebo. Participants have an equal chance of being assigned to either of the groups. For people that qualify and decide to participate in this study, they will be asked to make five visits to the study clinic and complete two study related phone calls over the course of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of autosomal dominant polycystic kidney disease (ADPKD).
* Estimated glomerular filtration rate (eGFR) > 50 ml/min/1.73m2 as determined from the serum creatinine by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Provide Informed consent

Exclusion Criteria:

* History of liver disease or abnormal liver function test
* Heavy alcohol intake
* Chronic diarrhea or malabsorption syndrome
* Thrombocytopenia
* Hypophosphatemia
* Pregnancy or lactation or plan to become pregnant during the study
* Treatment with anti-epileptic drugs
* Treatment with tolvaptan, current or within 2 months prior to screening
* Participation in another interventional trial currently or within 2 months prior to screening.

Exclusions specific to magnetic resonance (MR) imaging acquisition and measurement:

* Partial or total nephrectomy or renal cyst reduction (including aspiration) done <1 year ago
* Cardiac pacemaker.
* Presence of MR incompatible metallic clips (e.g. clipped cerebral aneurysm)
* Body weight >159 kg (350 lbs) or untreatable claustrophobia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Change in acetylated/total p53 ratio measured by ELISA in peripheral blood mononuclear cells (PBMC) | Change from Baseline to Month 12
  Sirtuin 1 deacetylates p53 protein, and niacinamide inhibits sirtuin 1. So an increase in acetylated/total p53 ratio in PBMC will be used as a marker of biological efficacy.

SECONDARY OUTCOMES:
Change in height-adjusted total kidney volume | Change from Baseline to Month 12
  Measured by MRI
Change in score on pain questionnaire | Change from Baseline to Month 12
  PKD-9 Pain Questionnaire: Range of scores from 13 (no pain or symptoms) to 70 (very severe symptoms almost every day)
Change in urinary concentration of MCP-1 | Change from Baseline to Month 12
Change in estimated GFR | Change from Baseline to Month 12
  Determined from serum creatinine concentrations using CKD-Epi equation

CONTACTS AND LOCATIONS:
Overall Officials: Alan Yu, M.B., B.Chir, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039